CLINICAL TRIAL: NCT05907109
Title: NeuroCardio Baby Research Outpatient Clinic: Study on the Neurodevelopment of Infants With Congenital Heart Disease in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Lucchese, PHD, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4864543
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Congenital Heart Disease; Child Development; Early Intervention
Keywords: Congenital Heart Disease; Child Development; Early Intervention; Telemonitoring; Home-based intervention
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Prospective Multicentric single-blinded, Two-arm Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Assessors blinded to the allocation of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Remotely monitored parent-mediated hybrid home and clinic based multidisciplinary Early Intervention protocols.
  Interventions: Behavioral: Remotely monitored parent-mediated hybrid home and clinic based multidisciplinary Early Intervention protocols.
- Control Group - Standart of Care (No Intervention): * The control group receives basic guidelines on child development, nutrition, and breastfeeding provided by the Brazilian Ministry of Health, in addition to standard of care cardiac pediatric follow-up visits.
  * Infants will receive outcome developmental evaluations within a 42-month follow-up clinic.

INTERVENTIONS:
Behavioral: Remotely monitored parent-mediated hybrid home and clinic based multidisciplinary Early Intervention protocols. — * Parents receive manualized protocols, instructional videos, and toy and material kits to administer EIs at home.
  * New modules are provided according to infant age or stage of intervention during the length of brief interventions or 12-months.
  * The families will be monitored by clinical researchers weekly. -High risk infants will receive supplemental EI services at the clinic according to developmental needs.
  * Infants will receive outcome evaluations within a 42-month follow-up clinic.
  Arms: Intervention

SUMMARY:
The objective of this randomized clinical trial is to test the effectiveness of a low-cost hybrid remotely monitored parent-mediated and clinic-based multidisciplinary early intervention (EI) for low-income infants with CHD in Brazil. The intervention protocols will be administered according to age modules, families will be monitored weekly. High risk infants also receive supplemental clinic-based interventions according to developmental needs. Controls will receive standard of care and access to early child development and nutrition practices information from the Brazilian Ministry of Health. All infants will be evaluated at within a 42-month follow-up research outpatient clinic, called NeuroCardio Baby at Santo Antonio Pediatric Hospital, of the Santa Casa de Misericordia Hospital Complex, and affiliated with The Cardiology Institute-University Foundation of Cardiology (IC-FUC), Porto Alegre, Brazil.

DETAILED DESCRIPTION:
The objective of this randomized clinical trial is to develop low-cost hybrid remotely monitored parent-mediated multidisciplinary early intervention (EI) protocols for infants with CHD in Brazil. The protocols will be conducted via parents at home according to age modules (0- 3m, 3-6m, 6-9m, and 9-12m), and families will be monitored by clinical researchers weekly. High risk infants will receive supplemental EI services at the clinic according to developmental needs. Infants will receive outcome evaluations within a 42-month follow-up clinic. The aim of this study is to prevent or reduce neurodevelopmental sequelae and developmental delays associated with CHD. Participants in the intervention group receive multidisciplinary EIs in Nutrition (including breastfeeding support), Speech and Language Therapy for tube feeding transition, feeding readiness, and language and motor development and early stimulation for global development in cognitive, language and motor skills according to age milestones. Premature infants will receive age-corrected protocols and evaluations. Caregivers will receive psychological and protocol administration support. The control group receives basic child development, nutrition, and breastfeeding information provided by the Brazilian Ministry of Health, in addition to standard of care cardiac pediatric follow-up visits. Neurodevelopment is assessed with the Brazilian Version of Bayley Developmental Scale for Infants and Toddlers (3rd edition) in both groups, at 6, 12, 24, and 36-42 months. Nutritional outcomes, such as ml of breastmilk drown by mothers, and infant weight and length are measured. The study will compare the developmental outcome scores and parental quality of life scores of the intervention and control groups during the intervention (6 and 12months) and at 1 and 2 years follow up. We believe that infants with CHD who receive monitoring and early multidisciplinary interventions in the first year of life have better neurodevelopmental outcomes than infants who do not receive early multidisciplinary care. In Brazil, access to EI services is extremely limited to urban centers and higher income families. Infants from low-income backgrounds and rural settings are likely to be left without services during early childhood. Our remote, low-cost intervention aims at increasing access to EI for Brazilian infants with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a fetal diagnosis of CHD
* Child up to two months diagnosed with CHD
* Signature of the electronic free and informed consent form by those parents or legal guardians.

Exclusion Criteria:

* Psychiatric or neurocognitive condition that prevents obtaining reliable clinical data (defined by the clinical judgment of the investigators)
* Inability to read by parents or legal guardians.

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compose the Neuropsychomotor profile of babies with CHD in multidisciplinary outpatient follow-up and compare to the group without follow-up. | From six months of age
  Compose the Neuropsychomotor profile of babies with CHD in multidisciplinary outpatient follow-up and compare to the group without follow-up using Bayley Scales of Infant and Toddler Development- Third Edition).

SECONDARY OUTCOMES:
Neurodevelopment Scores in infant with CHD (Bayley Scales of Infant and Toddler Development- Third Edition) | From six months of age
  Amercian Heart Association recommends surveillance, screening, evaluation in the nerudovelopment in pediatric congenital heart disease (CHD) population. The Bayley Scales of Infant and Toddler Development- Third Edition is a recognized scale the assessment the Infant Neudevelopment in cognitive, language and motor domains.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lucchese-Lobato, PHD, Principal Investigator — Instituto De Cardiologia/Fundação Universitária De Cardiologia
Locations (2):
- Brazil (2):
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Result] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541
- [Derived] Michelon RC, Lucchese-Lobato F. A remote parent-led early intervention protocol to promote motor development in infants with congenital heart disease: a feasibility pilot study of a randomized clinical trial. Dev Neurorehabil. 2024 Apr-May;27(3-4):134-144. doi: 10.1080/17518423.2024.2365796. Epub 2024 Jun 26. PMID 38922306
- See also: Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association — https://pubmed.ncbi.nlm.nih.gov/22851541/